CLINICAL TRIAL: NCT03707301
Title: Post-SOPHrology Cancer Patients' anxieTY Report
Acronym: SOPHTY
Status: Terminated | Type: Observational
Why Stopped: Enrollment difficulties
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-0203; 2018-A02004-51 (Other: ANSM)
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Cancer
Keywords: Cancer; Sophrology; Anxiety; Hospital Anxiety and Depression scale
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patients performing sophrology sessions: Cancer patients performing sophrology sessions will be recruited in this study, and will complete questionnaires of satisfaction and the Hospital Anxiety and Depression scale.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Questionnaires of satisfaction and the Hospital Anxiety and Depression scale.

SUMMARY:
Cancer is pathology with a high impact on patients and relatives quality of life. Most of the time, it is a stressful trial. Professionals have often resort to pharmaceutical solutions, but sometimes, it is not sufficient. So, patients resort to alternative and complementary medicines, as sophrology. In Lucien Neuwirth Cancer Institute, patients can benefit from sophrology.

Anxiety levels have never been reported before and after sessions. Indeed, the present study wants to report anxiety levels before, after, and one and three weeks after session. Levels of satisfaction will also be reported.

DETAILED DESCRIPTION:
Cancer is pathology with a high impact on patients and relatives quality of life. Most of the time, it is a stressful trial. Professionals have often resort to pharmaceutical solutions, but sometimes, it is not sufficient. So, patients resort to alternative and complementary medicines, as sophrology. In Lucien Neuwirth Cancer Institute, patients can benefit from sophrology.

Anxiety levels have never been reported before and after sessions. Indeed, the present study wants to report anxiety levels before, after, and one and three weeks after session. Levels of satisfaction will also be reported.

ELIGIBILITY:
Inclusion Criteria:

- Patient performing at least one session of sophrology in the Lucien Neuwirth Cancer Institute

Exclusion Criteria:

* Protected patient (according to the law),
* Patient with incapacity to complete questionnaires,
* Patient with incapacity to perform sophrologic movements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients performing sophrology sessions at the Lucien Neuwirth Cancer Institute will be recuited in this study.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Level of anxiety difference | 1 hour
  Level of anxiety after sophrology session will be compared to the level of anxiety before session, on a visual scale from 0 to 10. The scale is 10 centimeters long, printed on a paper.

SECONDARY OUTCOMES:
Level of anxiety difference | 1 month
  Level of anxiety after a second session of sophrology will be compared to the level of anxiety reported before the first sophrology session, according to the Hospital Anxiety and Depression scale, part A. The part A is composed of seven questions, with a score obtained between 0 and 28. A score between :
  * 7 or less : no symptomatology ;
  * 8 to 10 : doubtful symptomatology ;
  * 11 and more : certain symptomatology.
Level of depression difference | 1 month
  Level of depression after a second session of sophrology will be compared to the level of depression reported before the first sophrology session, according to the Hospital Anxiety and Depression scale, part B. The part B is composed of seven questions, with a score obtained between 0 and 28. A score between :
  * 7 or less : no symptomatology ;
  * 8 to 10 : doubtful symptomatology ;
  * 11 and more : certain symptomatology.
Sessions duration | 1 hour
  Duration of sessions will be reported, unit used: minutes.
Number of sessions | 1 month
  Number of sessions performed during one month will be reported.
Patients satisfaction | 1 month
  Patients satisfaction will be reported during one month, as many times as they performed sophrology sessions, on a visual scale from 0 to 10. The scale is 10 centimeters long, printed on a paper.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Morisson, MD, Principal Investigator — Institut de Cancérologie Lucien Neuwirth
Locations (1):
- Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez, France

IPD SHARING:
Plan to Share IPD: No